CLINICAL TRIAL: NCT00725530
Title: Evaluation of Deposits on Contact Lenses Worn Extended Wear
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Alcon Research (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single
Other Study IDs: MS-007
Record Dates: First submitted 2008-07-28; First posted 2008-07-30 (Estimated); Results first posted 2012-08-22 (Estimated); Last update posted 2012-08-22 (Estimated); Status verified 2012-07

CONDITIONS: Myopia
Keywords: Lens deposits; Soft contact lens wearers
MeSH Terms: conditions — Myopia

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- balafilcon A / etafilcon A (Active Comparator): Balafilcon A worn first, with etafilcon A worn second. Each product worn bilaterally in an extended wear (overnight) basis for 7 days.
  Interventions: Device: balafilcon A contact lens (PureVision); Device: etafilcon A contact lens (Acuvue2)
- etafilcon A / balafilcon A (Active Comparator): Etafilcon A worn first, with balafilcon A worn second. Each product worn bilaterally in an extended wear (overnight) basis for 7 days.
  Interventions: Device: balafilcon A contact lens (PureVision); Device: etafilcon A contact lens (Acuvue2)

INTERVENTIONS:
Device: balafilcon A contact lens (PureVision) — Commercially marketed, silicone hydrogel contact lens
  Other Names: PureVision
Device: etafilcon A contact lens (Acuvue2) — Commercially marketed, hydrogel contact lens
  Other Names: Acuvue2

SUMMARY:
The purpose of this study was to measure lipid deposits on commercially marketed contact lenses when worn on an extended wear (overnight) basis for 7 days.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 or older.
* Visual acuity correctable to 20/30 (Snellen) or better in each eye at distance with contact lenses.
* Successfully wearing hydrogel or silicone hydrogel contact lenses.
* Other protocol-defined inclusion criteria may apply.

Exclusion Criteria:

* Evidence or history of ocular conditions as prescribed in the protocol.
* One functional eye or a monofit lens.
* Any slit-lamp finding score of (1) at the Screening Visit as defined by the protocol.
* Use of concomitant topical ocular prescription or over-the-counter ocular medications.
* History of seasonal allergies with significant ocular side effects.
* Other protocol-defined exclusion criteria may apply.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 54 (Actual)
Dates: Start 2008-03; Primary Completion 2008-10 (Actual); Study Completion 2008-10 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Alcon Call Center for Trial Locations, Fort Worth, Texas, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Each site enrolled normal participants (non-depositors) and depositors in approximately a 1:1 ratio, as outlined in the protocol. 54 participants in 3 US sites and 1 UK site were enrolled.
Pre-assignment Details: Participants meeting eligibility criteria at the screening visit were enrolled into the study. 48 hours of no lens wear prior to Visit 1 served as the washout period. This reporting group includes all enrolled and dispensed participants.
Period: First Intervention, 7 Days (+0/-1)
Arm/Group | Balafilcon A / Etafilcon A | Etafilcon A / Balafilcon A
Started | 27 | 27
Completed | 27 | 27
Not Completed | 0 | 0
Period: Second Intervention, 7 Days (+0/-1)
Arm/Group | Balafilcon A / Etafilcon A | Etafilcon A / Balafilcon A
Started | 27 | 27
Completed | 27 | 27
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Overall: This reporting group includes all enrolled and dispensed participants.
Arm/Group | Overall
Number analyzed (Participants) | 54
Age Continuous [Mean (Standard Deviation); unit: years] | 32.35 (12.71)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 42
  Male | 12

OUTCOME MEASURES:

1. Primary Outcome: Front Surface Lens Deposits
Description: Film and discrete deposits were assessed with a slit-lamp after 2-5 hours of open eye lens wear. Film deposits were recorded on a 5-point scale, where 0=no deposition, clean surface; 1=slight, deposition occupying 1-5% of lens front surface; 2=mild, deposition occupying 6-15% of lens front surface; 3=moderate, deposition occupying 16-25% of lens front surface; 4=severe, deposition occupying >25% of lens front surface. Discrete deposits were recorded on a 5-point scale, where 0=no deposition, clean surface; 1=microdeposits (less than or equal to 10 dots); 2=microdeposits (greater than 10 dots); 3=macro deposits; 4=one or more jelly bumps. Participants were classified into Front Surface Lens Deposits <2 (less than grade 2 for both film and discrete) and into front surface lens deposits >1 (greater than grade 1 for either film, discrete, or both).
Time Frame: 7 days
Population: All enrolled participants.
Measure: Number; unit: Participants
Groups:
- Balafilcon A: Commercially marketed, silicone hydrogel, soft contact lenses worn for 7 days on an extended wear (overnight) basis.
- Etafilcon A: Commercially marketed, hydrogel, soft contact lenses worn for 7 days on an extended wear (overnight) basis.
Arm/Group | Balafilcon A | Etafilcon A
Number analyzed (Participants) | 54 | 54
Participants
  Deposits graded <2 | 20 | 25
  Deposits graded >1 | 34 | 29

ADVERSE EVENTS:
Time Frame: Adverse events were collected for the duration of the study.
Description: Safety data was collected on all enrolled and dispensed participants.
Groups:
- Balafilcon A Contact Lenses: Commercially marketed, silicone hydrogel, soft contact lenses worn for 7 days on an extended wear (overnight) basis.
Arm/Group | Balafilcon A Contact Lenses | Etafilcon A
Serious Adverse Events (participants affected / at risk) | 0/54 | 0/54
Other Adverse Events (participants affected / at risk) | 0/54 | 0/54

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less